CLINICAL TRIAL: NCT06072833
Title: Characterizing and Addressing Financial Toxicity in Adolescents and Young Adults With Cancer
Brief Title: Characterizing and Addressing Financial Toxicity in AYAs With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Patient Advocate Foundation (Unknown); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Melissa Beauchemin, Assistant Professor of Nursing, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAU2405; 5KL2TR001874 (NIH)
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Cancer in Adolescence
Keywords: Cancer; Adolescents; Young Adults; Financial Needs; Social Needs; Minority health; Caregivers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants who screen positive all move forward to receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient Financial Education / Navigation (Experimental): Individuals who screen positive will all move forward to receive the intervention. This intervention includes partnering with community-based organizations to deliver financial education, connection to resources, and counseling tailored to individual patients and spouses for 6-months.
  Interventions: Behavioral: Patient Financial Education / Navigation

INTERVENTIONS:
Behavioral: Patient Financial Education / Navigation — The investigator anticipates that this will include a baseline financial assessment and educational content, likely using a virtual platform. Participants will be connected with a PAF case manager. There will be monthly follow-ups to the participant for 6-months to address any financial concerns through additional counseling/navigation.

SUMMARY:
The overall aims of this study are to address two important gaps in care for AYA cancer patients: 1) a financial toxicity measurement tool to assess AYA-specific needs, and 2) an intervention for mitigating financial toxicity in this population. Aim 1 involves adapting the COSTA measure and assessing the psychometric properties of the measure for a racial/ethnically diverse group of AYAs. Aim 2 and 3 involve the development and pilot testing of our novel financial education/ navigation (FE/FN) intervention.

DETAILED DESCRIPTION:
Financial toxicity is the harmful personal financial burden faced by patients due to healthcare needs. A prevalent adverse outcome of cancer therapy, financial toxicity is associated with poorer health outcomes and increased mortality in adults with cancer. Among cancer survivors, financial burden disproportionately impacts adolescents and young adults (AYA: 15 - 39 years). Lack of financial security, insurance gaps or under-insurance, and interruptions in education or careers caused by cancer therapy make AYA cancer survivors particularly vulnerable to financial burden. Financial toxicity of cancer care is an actionable factor impacting outcomes among vulnerable AYA populations. In order to improve outcomes and reduce the burden of care among these populations, targeted, appropriate measures and then, age-specific interventions are needed. The study includes the following aims: Aim 1 involves the adaptation of the COST measure and assessment of the psychometric properties of the measure for a racial/ethnically diverse group of AYAs. The study team will administer COST and additional AYA-specific financial toxicity candidate items to N=150 AYAs. The study will assess validity of original COST through confirmatory factor analysis; assess reliability through test/retest; conduct exploratory factor analysis on modified COST incorporating added items; and describe AYA-reported acceptability of AYA financial toxicity assessment.

In Aim 2, an adapted FN/FE intervention will be adapted for a racial/ethnically diverse group of AYAs. 6 focus groups (6 - 8 per group) will be conducted with a diverse AYAs and caregivers, and brief stakeholder discussions to understand unique AYA FE/FN needs and inform intervention refinement.

Aim 3 will include a pilot test of our novel FE/FN intervention to AYAs. A FE/FN intervention will be delivered to at least N=30 AYAs, and assess feasibility by evaluating program completion (6-months), participant-reported acceptability. Evidence of efficacy will be recorded by measuring improvement in average financial toxicity score between baseline and 6-month time points.

ELIGIBILITY:
Inclusion Criteria:

AYA patient participants:

* Age 15 - 39 years old
* English or Spanish-speaking
* Diagnosed with cancer that required treatment within past 18 months
* Not currently on hospice care

Caregiver/financial partner participants:

* Parent or financially-responsible adult of non-adult AYA (<18 years) OR
* Identified by the AYA as caregiver, parent, or partner who is financially-responsible or a financial partner for AYA

Exclusion Criteria:

* Unable to complete financial survey questions or contraindicated (as outlined in Protection of Human Subjects)

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Number of (OR percentage of) participants who completed the intervention | Up to 6 months
  This is to assess the feasibility of intervention completion. Intervention completion is defined as participants who have demonstrated contact with community partners at any time before the end of 6 months.
Percentage of eligible participants who consented to be in study | Up to 6 months
  This is to measure interest and the need for help by community partners that can provide patient financial education and navigation.

SECONDARY OUTCOMES:
Comprehensive Score of Financial Toxicity (COST measure) | Baseline, 6 months
  The COST is a patient-reported outcome measure that describes the financial distress experienced by cancer patients. It is a 11-item questionnaire with a score range of 0-44. Lower COST values indicate higher toxicity. Higher scores indicate lower financial toxicity .

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Beauchemin, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zafar SY, Peppercorn JM, Schrag D, Taylor DH, Goetzinger AM, Zhong X, Abernethy AP. The financial toxicity of cancer treatment: a pilot study assessing out-of-pocket expenses and the insured cancer patient's experience. Oncologist. 2013;18(4):381-90. doi: 10.1634/theoncologist.2012-0279. Epub 2013 Feb 26. PMID 23442307
- [Background] Altice CK, Banegas MP, Tucker-Seeley RD, Yabroff KR. Financial Hardships Experienced by Cancer Survivors: A Systematic Review. J Natl Cancer Inst. 2016 Oct 20;109(2):djw205. doi: 10.1093/jnci/djw205. Print 2017 Feb. PMID 27754926
- [Background] Yabroff KR, Dowling EC, Guy GP Jr, Banegas MP, Davidoff A, Han X, Virgo KS, McNeel TS, Chawla N, Blanch-Hartigan D, Kent EE, Li C, Rodriguez JL, de Moor JS, Zheng Z, Jemal A, Ekwueme DU. Financial Hardship Associated With Cancer in the United States: Findings From a Population-Based Sample of Adult Cancer Survivors. J Clin Oncol. 2016 Jan 20;34(3):259-67. doi: 10.1200/JCO.2015.62.0468. Epub 2015 Dec 7. PMID 26644532
- [Background] Parsons HM, Harlan LC, Lynch CF, Hamilton AS, Wu XC, Kato I, Schwartz SM, Smith AW, Keel G, Keegan TH. Impact of cancer on work and education among adolescent and young adult cancer survivors. J Clin Oncol. 2012 Jul 1;30(19):2393-400. doi: 10.1200/JCO.2011.39.6333. Epub 2012 May 21. PMID 22614977
- [Background] Nipp RD, Kirchhoff AC, Fair D, Rabin J, Hyland KA, Kuhlthau K, Perez GK, Robison LL, Armstrong GT, Nathan PC, Oeffinger KC, Leisenring WM, Park ER. Financial Burden in Survivors of Childhood Cancer: A Report From the Childhood Cancer Survivor Study. J Clin Oncol. 2017 Oct 20;35(30):3474-3481. doi: 10.1200/JCO.2016.71.7066. Epub 2017 Aug 17. PMID 28817372
- [Background] de Souza JA, Yap BJ, Wroblewski K, Blinder V, Araujo FS, Hlubocky FJ, Nicholas LH, O'Connor JM, Brockstein B, Ratain MJ, Daugherty CK, Cella D. Measuring financial toxicity as a clinically relevant patient-reported outcome: The validation of the COmprehensive Score for financial Toxicity (COST). Cancer. 2017 Feb 1;123(3):476-484. doi: 10.1002/cncr.30369. Epub 2016 Oct 7. PMID 27716900
- [Background] Danhauer SC, Canzona M, Tucker-Seeley RD, Reeve BB, Nightingale CL, Howard DS, Puccinelli-Ortega N, Little-Greene D, Salsman JM. Stakeholder-informed conceptual framework for financial burden among adolescents and young adults with cancer. Psychooncology. 2022 Apr;31(4):597-605. doi: 10.1002/pon.5843. Epub 2021 Nov 5. PMID 34699110
- [Background] Beauchemin MP, Elkin EB, Wright JD, Kukafka R, Hershman DL, Kahn J. Incorporating systematic financial screening into the electronic health record. Journal of Clinical Oncology. 2021;39(28_suppl):184-184.
- [Derived] Khurana RK, Valera K, Raghunathan R, Gallagher KD, Angove RS, Bradshaw E, Patton J, Alvarado S, Crespo S, Judon K, DiCola K, Steinberg DM, Wang S, Hershman DL, Beauchemin MP. Pilot feasibility of a financial and health-related social needs navigation intervention (AYA-NAV) for adolescents and young adults with Cancer: Study protocol for a prospective, single-arm study. Contemp Clin Trials Commun. 2025 Jul 16;47:101523. doi: 10.1016/j.conctc.2025.101523. eCollection 2025 Oct. PMID 40726516